CLINICAL TRIAL: NCT04474080
Title: The Role of Virtual Peer Support Platforms for Reducing Stress and Burnout Among Frontline Healthcare Workers During COVID-19: a Pilot Randomized Controlled Trial
Brief Title: Reducing Burnout Among Frontline Healthcare Workers During COVID-19
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Zainab Samaan (Zena), Associate Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 11136
Record Dates: First submitted 2020-07-08; First posted 2020-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Burnout
Keywords: physician; burnout; COVID-19; public health response; stress; depression; virtual peer support platforms; frontline healthcare workers
MeSH Terms: conditions — Burnout, Psychological; COVID-19; Depression

STUDY DESIGN:
Intervention Model Description: The following trial uses a nested stepped-wedge randomized controlled trial design. Specialty residency programs will be the unit of randomization, with each program being randomized to receive the virtual peer support intervention across varying time-points. An in-depth evaluation of the interventions acceptability will be completed using a nested qualitative study design, wherein a subgroup of participants (preferably across residency programs) will be invited to participate in a brief 10-minute interview to explore their experiences with the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Peer Support Platform (Experimental): The intervention program content will be informed by "the BASICS"-a guide for supporting resilience against burnout, developed by the Ontario Medical Association Physician Health Program, as well as the Person-Environment-Occupation (PEO) model, a transactive approach to modelling occupational performance issues in the field of Occupational Therapy. "The BASICS" highlights six fundamental domains will underlie the focus of group therapy sessions, where participants will be encouraged to consider how they may incorporate healthy physical and emotional practices both on their own (Person), and during the practice of medicine (Occupation), in addition to identifying barriers to adopting these practices within the healthcare environment (Environment).
  Interventions: Behavioral: Virtual Peer Support Platform
- Control period (Active Comparator): Residents will continue with their regular academic day activities during the allotted intervention time.
  Interventions: Behavioral: Control Period

INTERVENTIONS:
Behavioral: Virtual Peer Support Platform — The intervention program will consist of 6 virtual 30-minute sessions delivered across three months. Sessions will follow a structured format including: check-in, issue identification & context, facilitated discussion, environmental strategies, occupational strategies, experiential component, as well as summary and sign-out. Meetings will finish with a stress relieving activity, to be performed together on the web-based platform. The facilitated discussions will follow important themes including focus on self, patients, and external stressors.
  Arms: Virtual Peer Support Platform
Behavioral: Control Period — The control period will be the time prior to randomization and commencement of the intervention, whereby residents will continue with their regular academic day activities during the allotted intervention time
  Arms: Control period

SUMMARY:
Physician burnout has a significant impact on the wellness and productivity of physicians as well as patient health outcomes. Managing burnout among frontline workers is critical to Canada's response to the COVID-19 pandemic, in order to support frontline workers and reduce inefficiencies and medical errors frequently linked to burnout, ultimately improving our ability to detect, treat and manage COVID-19 cases. Therefore, this trial aims to assess the effects of an 8-session intervention over 3 months for burnout in physician residents in residency programs at McMaster University in Canada during the COVID-19 pandemic. This trial will provide evidence to inform health system management and public health response early and effectively so as to maintain the integrity of our workforce during and post-pandemic. The virtual delivery platform renders the proposed intervention easily disseminated internationally, in low- middle- and high- income countries and across urban and rural cities.

DETAILED DESCRIPTION:
Physician burnout has come to the forefront of discourse within the medical field due to its significant impact on the wellness and productivity of physicians as well as patient health outcomes. Burnout is defined as physical, mental and emotional exhaustion resulting from persistent exposure to an emotionally demanding trigger, and is comprised of three dimensions: emotional exhaustion (EE), depersonalization (DP) and lack of personal accomplishment (PA). Residency is a particularly stressful time; the junior physician is tasked with a tremendous responsibility of providing high quality care while learning and integrating new skills during training. Adapting to these job demands has a direct consequence on one's emotional reserve and ability to establish a healthy home-work interface. Recent data indicates 47% of residents around the world suffer from burnout, and that rates are highest in North America.

During times of lethal pandemics, healthcare workers (HCWs) have a duty to serve on the frontline. Within three months of the first report of COVID-19, a global pandemic was declared and social separation and economic shutdowns were enforced around the globe. Meanwhile, resident physicians were redeployed to the frontline by their training institutions, inevitably jeopardizing their speciality training. In addition to the detrimental personal and substantial financial stressors generally incurred by persons during a pandemic, residents bear the burden of caring for others and witnessing tragic outcomes thus putting them at risk of "accelerated burnout". HCWs on the frontline during times of crisis and natural disaster historically suffer from more severe emotional distress, depression, anxiety, and social isolation. This is consistent with findings from a recent study of frontline workers in Wuhan, China during the COVID-19 pandemic, and reports of suicide among frontline workers attributed to COVID-19 associated stressors.

Many studies have aimed to delineate contributors of burnout and common themes that have emerged include excessive workloads, feeling unsupported, lack of autonomy, and lack of work-home integration. In addition to traditional causes of burnout, the heightened risk of occupational exposure to infection, process inefficiencies, limited resources, and financial instability have been established as additional stressors among HCWs during COVID-19. These factors, in addition to social stigmatization and ostracism by family and the fearful public have also been cited as major contributors to stress among HCWs during the Severe Acute Respiratory Syndrome (SARS) pandemic, the Ebola epidemic, and among HCWs caring for AIDS patients during the late 1980s.

Addressing burnout among frontline workers is essential to supporting Canada's response to the COVID-19 pandemic, in order to 1) keep our frontline workers on the frontline, and 2) reduce inefficiencies and medical errors frequently linked to burnout, ultimately improving our ability to detect, treat and manage COVID-19 cases. Based on evidence from previous pandemics, the investigators anticipate the grave impact of the pandemic on frontline workers will outlive the pandemic itself, and HCWs will continue to struggle with post-traumatic stress in the midst of a crashing economy and more than ever strained healthcare system. To address this serious threat to health workers globally, the investigators wish to evaluate the effectiveness and acceptability of a virtual peer support program in reducing overall burnout among resident physicians during COVID-19 pandemic. Using an adapted intervention from West et. al, modified to six support sessions delivered across three months, the investigators will randomize different medical specialties to receiving this intervention employing a stepped wedged pilot randomized trial design. The goals of the pilot trial will be to assess feasibility of adapting an in-person group-based intervention to virtual platforms across multiple subspecialty residency programs at a single post-graduate medical education (PGME) institution in Ontario, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Physician residents across all medical specialties at McMaster University, McGill University, and Stanford University.
* Must be able to provide written informed consent

Exclusion Criteria:

* Residents who are on prolonged leave (>4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Acceptability as assessed through patient reported experiences with the virtual intervention. | Month 3
  Qualitative interviews to explore participants impressions and experiences with virtually adapted burnout intervention. A subgroup of participants (preferably across residency programs), will be invited to participate in a brief 10-minute interview to explore their experiences with the intervention through semi-structured open ended interview questions.
Recruitment | To be assessed at three months
  Total number of participants recruited to the study
Retention | To be assessed at the end of the observation period. The duration of the observation period will be based on the total number of residency programs enrolled in the study given the stepped-wedge design.
  Total number of participants who remain in the study until the end of observation
Number of sessions completed | To be assessed at the end of the three month intervention period.
  Measured as number of sessions completed
Average group size | To be assessed at the end of the three month intervention period.
  Measured as the mean number of participants per group
Data completion | To be assessed at the end of the three month intervention period
  Measured as the percentage of instruments completed
Feasibility of adapting an in-person group-based intervention to virtual platforms as assessed by group participation rates and self-reported experiences with the intervention. | To be assessed at the end of the three month intervention period.
  Feasibility will be assessed by evaluation of 1) participation rates across the intervention period, and 2) self-reported feedback about experiences with the intervention as gathered through survey responses. Survey questions will specifically ask about user experience with the intervention materials, technology including virtual platform.

SECONDARY OUTCOMES:
Assess stress | This is not a time to event variable. We will be evaluating the change from baseline and three months post initiation of intervention
  Instrument/method of measurement: Stress will be measured using the Perceived Stress Scale, a 10-item scale ranging from 0-4 representing never to very often, with total scores between 0-40.
Assess depression | This is not a time to event variable. We will be evaluating the change from baseline and three months post initiation of intervention
  Instrument/method of measurement: Depression will be measured using a feasible two question approach developed by Spitzer et. al, validated by Whooley et. al.
Quality of life as assessed by a validated single item linear analogue scale. | This is not a time to event variable. We will be evaluating the change from baseline and three months post initiation of intervention
  Instrument/method of measurement: Single item linear analog scale. A score of 5 or less on this scale has known association with poor outcomes across clinical research of burnout.
Assess and measure overall burnout | This is not a time to event variable. We will be evaluating the change from baseline and three months post initiation of intervention.
  Instrument/method of measurement: Maslach Burnout Inventory (MBI) will be administered to measure overall burnout. The MBI is a 22-item measure of the three dimensions of burnout: emotional exhaustion (EE), depersonalization (DP) and lack of personal accomplishment (PA) on a 7-point Likert scale ranging from 0 to 6. High scores on EE (≥26) or DP (≥9), and low scores on PA (≤34) are indicative of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Samaan, MBChB, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zis P, Anagnostopoulos F, Sykioti P. Burnout in medical residents: a study based on the job demands-resources model. ScientificWorldJournal. 2014;2014:673279. doi: 10.1155/2014/673279. Epub 2014 Oct 30. PMID 25531003
- [Background] Grobler L, Mehtar S, Dheda K, Adams S, Babatunde S, van der Walt M, Osman M. The epidemiology of tuberculosis in health care workers in South Africa: a systematic review. BMC Health Serv Res. 2016 Aug 20;16(1):416. doi: 10.1186/s12913-016-1601-5. PMID 27544429
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Montemurro N. The emotional impact of COVID-19: From medical staff to common people. Brain Behav Immun. 2020 Jul;87:23-24. doi: 10.1016/j.bbi.2020.03.032. Epub 2020 Mar 30. No abstract available. PMID 32240766
- [Background] Ishak W, Nikravesh R, Lederer S, Perry R, Ogunyemi D, Bernstein C. Burnout in medical students: a systematic review. Clin Teach. 2013 Aug;10(4):242-5. doi: 10.1111/tct.12014. PMID 23834570
- [Background] Thomas NK. Resident burnout. JAMA. 2004 Dec 15;292(23):2880-9. doi: 10.1001/jama.292.23.2880. PMID 15598920
- [Background] Sasangohar F, Jones SL, Masud FN, Vahidy FS, Kash BA. Provider Burnout and Fatigue During the COVID-19 Pandemic: Lessons Learned From a High-Volume Intensive Care Unit. Anesth Analg. 2020 Jul;131(1):106-111. doi: 10.1213/ANE.0000000000004866. No abstract available. PMID 32282389
- [Background] Shiao JS, Koh D, Lo LH, Lim MK, Guo YL. Factors predicting nurses' consideration of leaving their job during the SARS outbreak. Nurs Ethics. 2007 Jan;14(1):5-17. doi: 10.1177/0969733007071350. PMID 17334166
- [Background] Koh D, Lim MK, Chia SE, Ko SM, Qian F, Ng V, Tan BH, Wong KS, Chew WM, Tang HK, Ng W, Muttakin Z, Emmanuel S, Fong NP, Koh G, Kwa CT, Tan KB, Fones C. Risk perception and impact of Severe Acute Respiratory Syndrome (SARS) on work and personal lives of healthcare workers in Singapore: what can we learn? Med Care. 2005 Jul;43(7):676-82. doi: 10.1097/01.mlr.0000167181.36730.cc. PMID 15970782
- [Background] Li Y, Wang H, Jin XR, Li X, Pender M, Song CP, Tang SL, Cao J, Wu H, Wang YG. Experiences and challenges in the health protection of medical teams in the Chinese Ebola treatment center, Liberia: a qualitative study. Infect Dis Poverty. 2018 Aug 16;7(1):92. doi: 10.1186/s40249-018-0468-6. PMID 30134982
- [Background] Barbour RS. Responding to a challenge: nursing care and AIDS. Int J Nurs Stud. 1995 Jun;32(3):213-23. doi: 10.1016/0020-7489(95)00003-g. PMID 7665310
- [Background] Whooley MA, Avins AL, Miranda J, Browner WS. Case-finding instruments for depression. Two questions are as good as many. J Gen Intern Med. 1997 Jul;12(7):439-45. doi: 10.1046/j.1525-1497.1997.00076.x. PMID 9229283
- [Background] Spitzer RL, Williams JB, Kroenke K, Linzer M, deGruy FV 3rd, Hahn SR, Brody D, Johnson JG. Utility of a new procedure for diagnosing mental disorders in primary care. The PRIME-MD 1000 study. JAMA. 1994 Dec 14;272(22):1749-56. PMID 7966923